CLINICAL TRIAL: NCT03990597
Title: A Pilot Study of StrataXRT, a Topical Silicone Barrier, to Prevent Auricular Radiation Dermatitis in Pediatric Patients Undergoing Proton Cerebrospinal Radiation Therapy
Brief Title: StrataXRT in Preventing Radiation Dermatitis in Pediatric Patients Undergoing Radiation Therapy to the Brain or Spinal Cord
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Per PI
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0980; NCI-2019-02709 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0980 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2020-11

CONDITIONS: Central Nervous System Sarcoma; Ependymoma; Glioma; Malignant Intracranial Germ Cell Tumor; Medulloblastoma; Pineoblastoma; Primary Central Nervous System Neoplasm
MeSH Terms: conditions — Ependymoma; Glioma; Medulloblastoma; Pinealoma; Central Nervous System Neoplasms | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Supportive care (StrataXRT, placebo) (Experimental): Beginning first day of CSI proton radiation therapy, caregivers apply StrataXRT gel to half of the patient's forehead and one ear and placebo to the other half of the forehead and the other ear BID until the last day of radiation therapy.
  Interventions: Other: Placebo Administration; Other: Questionnaire Administration; Drug: Wound Dressing Material

INTERVENTIONS:
Other: Placebo Administration — Applied topically
  Other Names: placebo; placebo therapy; PLCB; sham therapy
Other: Questionnaire Administration — Ancillary studies
Drug: Wound Dressing Material — Applied StrataXRT topically
  Other Names: Wound Dressing

SUMMARY:
This phase I trial studies the side effects of a silicone topical wound dressing (StrataXRT) and to see how well it works in preventing radiation dermatitis (skin burns and side effects caused by radiation) in pediatric patients undergoing radiation therapy. StrataXRT may help prevent or decrease severe skin rash, pain, itching, skin peeling, and dry skin in pediatric patients undergoing radiation therapy to the brain or spinal cord.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the safety (defined using the Common Terminology Criteria for Adverse Events [CTCAE], version 5.0) of StrataXRT and placebo by assessing gel-associated toxicities among pediatric patients, aged 2-17 undergoing proton cerebrospinal irradiation (CSI) for central nervous system (CNS) tumors.

II. To estimate the efficacy of StrataXRT as a preventative agent for radiation-associated dermatitis among pediatric patients, aged 2-17 undergoing proton CSI for CNS tumors.

SECONDARY OBJECTIVES:

I. To explore the relationship between dosing and the efficacy of StrataXRT. II. To explore the relationship between the use of StrataXRT and parent-reported symptom experience, as measured by the Radiation-Induced Skin Reaction Assessment Scale (RISRAS).

III. To explore compliance with the application of treatment as documented in a study log by participants.

OUTLINE:

Beginning first day of CSI proton radiation therapy, caregivers apply StrataXRT gel to half of the patient's forehead and one ear and placebo to the other half of the forehead and the other ear twice daily (BID) until the last day of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between the ages of 2 years old and 17 years old
* Patients diagnosed with primary CNS tumors including medulloblastoma, pineoblastoma, ependymoma, intracranial germ cell, glioma or intracranial sarcoma who will be starting proton CSI
* Patients planned to receive at least 20 Gy CSI at 1.8 - 2.0 Gy per fraction
* Patients with an identified adult (aged 18 years or older caregiver)(familial or other) who consents to apply the StrataXRT and placebo twice a day for the duration of the study and complete the study instruments
* Informed consent by parents or legal guardian; consent documents will be translated with non-English speaking participants

Exclusion Criteria:

* Patients who have already started proton CSI treatment
* Patients receiving > 10 fractions photon therapy
* Patients with pre-existing dermal scarring, as determined by a clinical member of the study staff
* Patients who only have a primary caregiver who is a minor (e.g. mother under the age of 18)
* Patients planned to receive less than 20 Gy CSI at 1.8-2.0 Gy per fraction

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 weeks
  Graded per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Safety will be summarized with standard summary statistics by adverse event (AE), grade, relation, etc. using the CTCAE 5.0. All summaries will be calculated for each control and experimental forehead and ears.
StrataXRT as a preventative agent for radiation-associated dermatitis | Up to 6 weeks
  To estimate the efficacy of StrataXRT among pediatric patients.

SECONDARY OUTCOMES:
Dosing of StrataXRT | Up to 6 weeks
Parent-reported symptom experience | Up to 6 weeks
  Will be measured by the Radiation-Induced Skin Reaction Assessment Scale (RISRAS). The RISRAS Radiation-Induced Skin Reaction Assessment Scale will be summarized by control and experimental ears at each time point (baseline, 5 weekly treatment visits, and at treatment completion visit [last day of radiation therapy]).
Compliance | Up to 6 weeks
  As documented in a study log by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L McGovern, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT03990597/ICF_000.pdf